CLINICAL TRIAL: NCT01267669
Title: A Double Blind Randomized Placebo-Controlled Trial of Somatostatin in Association With Endoscopic Variceal Ligation (EVL) in Control of Acute Variceal Bleeding
Brief Title: A Trial of Somatostatin With Endoscopic Variceal Ligation (EVL) in Control of Acute Variceal Bleeding
Acronym: AVB-EVL+S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr S K Sarin, Department of Gastroenterology, G B Pant Hospital, New Delhi, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-PHT-01
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Acute Bleeding Esophageal Varices; Portal Hypertension; Cirrhosis
Keywords: Variceal bleeding; Endoscopic therapy; Band ligation; Somatostatin; Vasoactive drugs; Octreotide
MeSH Terms: conditions — Hypertension, Portal; Fibrosis | interventions — Somatostatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVL plus Somatostatin (Experimental): Emergency EVL plus Somatostatin (250 mcg/hr) infusion for 5 days
  Interventions: Drug: Somatostatin
- EVL plus Placebo (Placebo Comparator): Emergency EVL plus placebo infusion for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Somatostatin — Emergency EVL plus Somatostatin (250 mcg/hr) infusion for 5 days
  Other Names: Somatosan; Somastin
  Arms: EVL plus Somatostatin
Drug: Placebo — Emergency EVL plus placebo infusion for 5 days
  Arms: EVL plus Placebo

SUMMARY:
Background: Efficacy of endoscopic variceal sclerotherapy in achieving initial control of acute variceal bleeding and five-day haemostasis has been shown to significantly improve when vasoactive drug is added. However, there is limited data whether addition of somatostatin, to endoscopic variceal ligation (EVL) improves the efficacy of EVL.

Aim: To compare EVL plus somatostatin versus EVL plus placebo in control of acute variceal bleeding.

Patients and methods: Consecutive cirrhotic patients with acute variceal bleeding from esophageal varices were enrolled in the trial. After emergency EVL, patients were randomized to receive either somatostatin (250 mcg/hr) or placebo infusion. Primary endpoint was treatment failure within 5 days. Treatment failure was defined as fresh hematemesis ≥2 hour after start of therapy or death.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of portal hypertension
* Having hematemesis and/or melena within 24 hour prior to admission
* Source of bleeding should be esophageal varices

Exclusion Criteria:

* Non-cirrhotic cause of portal hypertension
* Age <12 or >75 years
* Hepatic encephalopathy grade 3 or 4
* Renal failure with serum creatinine >2 mg/dL
* Any evidence of bleeding from additional source apart from esophageal varices (like gastric varices, portal hypertensive gastropathy, erosions or ulcers including variceal ulcers)
* Patients already on vasoactive drugs like somatostatin or terlipressin during the current episode of bleeding
* Patients already received EVL or EST elsewhere during the current episode of bleeding prior to presenting to our hospital
* Patients with history of surgery for portal hypertension or TIPS
* Concomitant severe cardio-pulmonary disease
* Concomitant malignancy
* HVPG not possible within 24 hrs of presentation
* Patients refusing to participate in the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 5 days
  The primary endpoint was treatment failure, defined as the occurrence of any of the following within a period of 120 h (5 days) from the time of admission: (i) Fresh hematemesis ≥2 hr after EVL; or (ii) Death within 5 days.

SECONDARY OUTCOMES:
In-hospital mortality | During the same admission
  Death during the same admission to the hospital
Transfusion requirement | During hospital stay
  Amount of packed cell or FFP infusions received during the hospital stay
ICU stay in days | During the hospital stay
  Number of dys the patient spent in ICU
Drug-related adverse effects | 5 days
  Adverse effects due to somatostatin or placebo infusion

CONTACTS AND LOCATIONS:
Overall Officials: Shiv K Sarin, MD, DM, Principal Investigator — G B Pant Hospital
Locations (1):
- Department of Gastroenterology, G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kumar A, Jha SK, Mittal VV, Sharma P, Sharma BC, Sarin SK. Addition of Somatostatin After Successful Endoscopic Variceal Ligation Does not Prevent Early Rebleeding in Comparison to Placebo: A Double Blind Randomized Controlled Trial. J Clin Exp Hepatol. 2015 Sep;5(3):204-12. doi: 10.1016/j.jceh.2015.06.001. Epub 2015 Jun 16. PMID 26628838